CLINICAL TRIAL: NCT00312715
Title: Thyroid Hormone-Induced Lipolysis: An In Vivo Microdialysis Study
Brief Title: Thyroid and Fat Tissue Metabolism
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060133; 06-DK-0133
Record Dates: First submitted 2006-04-08; First posted 2006-04-10 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2014-07-08

CONDITIONS: Healthy Volunteers
Keywords: Deiodinase; Levothyroxine; Liothyronine; Lipid Metabolism; Healthy Volunteer; HV

SUMMARY:
This study will use a technique called microperfusion to examine how thyroid hormones are involved in fat metabolism. The thyroid gland produces two kinds of hormones: T3 and T4. Some of the T4 is changed to T3 in various organs after leaving the thyroid. The T3 stimulates the body to burn fat. People have different rates at which they can change T4 to T3, and this may lead to differences in body fat among different people.

Microperfusion is based on the exchange of substances across tiny holes of a small plastic tube called a "probe," which is inserted after numbing the skin over a fat pad. Through these openings, the fat pad is continuously rinsed with small amounts of fluid, and an exchange of substances occurs. The fluid drips from the other opening of the probe and is collected in a vial. Small amounts of study drugs are infused and the amount of substances released by the fat pad in response to them are measured.

Healthy normal volunteers 18 years of age and older may be eligible for this study. Candidates are screened with a medical history, physical examination and blood tests.

Participants undergo microperfusion. A needle is placed in an arm vein for collecting blood samples before and at the end of the experiment for measuring thyroid hormones and other substances in the blood. The skin over the fat pad next to the umbilicus (navel) is numbed and two microperfusion probes are inserted. A salt water solution is infused into the fat pad for one hour and the substances in the fluid are measured as the fluid leaves the fat pad. After 1 hour isoproterenol, a drug that aids in energy production by fat, is added to help determine the level of fat metabolism. After an additional hour small amounts of thyroid hormone are added to the fluid and samples are collected as they leave the body. Two catheters are inserted during each experiment. Small volumes of sterile fluid are circulated continuously in the tubing and samples are collected at regular intervals.

DETAILED DESCRIPTION:
This study will examine how two thyroid preparations, levothyroxine (T4) and liothyronine (T3), affect subcutaneous adipose tissue in normal subjects. Thyroid hormone plays an important role in the maintenance of energy metabolism. Specifically, hyperthyroidism is associated with weight loss via an increase in metabolic rate and lipolysis. While this phenomenon has been studied in vitro quite extensively, very little information is available on the local action of thyroid hormone on adipose tissue in vivo and, in particular, at the present no information is available on the role of peripheral conversion of thyroid hormone in subcutaneous adipose tissue. We thus propose to study the local action of thyroid hormones on adipose tissue using microdialysis, a minimally invasive technique that allows the serial determination of components of the extracellular fluid. The measurement of glycerol after correction for changes in blood flow will be used to evaluate the effects of the thyroid hormones on local lipolysis.

Healthy volunteers 18 years of age and older may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood tests. Subjects with hyperlipidemia, impaired glucose tolerance or diabetes and thyroid disease are not eligible for the participation in this study. Qualifying study participants undergo subcutaneous fat tissue microdialysis to assess the effects of T3 and T4 on the activity of fat tissue. The medications isoproterenol and T3 or T4 are injected in fat tissue under the skin of the abdomen, and fluid samples are collected from the area over a 6-12 hour period using the same small needle. Glycerol is then measured to study how the thyroid hormones affect fat metabolism. During this procedure a 10% glucose solution is infused through the catheter in the arm to limit lipolysis due to fasting. Four different sets of experiments are performed with different thyroid hormone doses and/or durations.

These experiments will provide new information on the role of thyroid hormone in the regulation of adipose tissue metabolism and will help in identifying new treatments for the management of obesity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years, male or female.
* Written informed consent.

EXCLUSION CRITERIA:

* Hypo- or hyper-thyroid (history or TSH greater than 5.0 and less than 0.4 miU/L)
* Blood pressure greater than 140/90 mmHg [17] or current antihypertensive therapy
* History of cardiovascular disease
* BMI less than or equal to 20 or greater than or equal to 30 Kg/m(2).
* Diabetes mellitus (serum glucose greater than or equal to 126 mg/dL).
* Hypercholesterolemia (serum levels greater than or equal to 240 mg/dL), hypertriglyceridemia (plasma levels greater than or equal to 220 mg/dL) and/or use of antilipemic therapy.
* Liver disease or ALT serum level greater than two fold the upper laboratory reference limit.
* Renal insufficiency or estimated creatinine clearance less than or equal to 50 mL/min (Cockcroft method).
* History of illicit drug or alcohol abuse within the last 5 years; current use of drugs (by history) or alcohol (CAGE greater than 3).
* Psychiatric conditions or behavior that would be incompatible with safe and successful participation in this study
* Current use of medications/dietary supplements/alternative therapies known to alter thyroid function.
* Allergy to ethanol, levothyroxine, liothyronine, isoproterenol, lidocaine.
* Pregnancy/breastfeeding.
* Current smoker

All subjects will be fully informed of the aim, nature, and risks of the study prior to giving written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-04-03; Study Completion 2014-07-08

CONTACTS AND LOCATIONS:
Overall Officials: Francesco S Celi, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Elks ML, Manganiello VC. Effects of thyroid hormone on regulation of lipolysis and adenosine 3',5'-monophosphate metabolism in 3T3-L1 adipocytes. Endocrinology. 1985 Sep;117(3):947-53. doi: 10.1210/endo-117-3-947. PMID 2410243
- [Background] Germack R, Starzec A, Perret GY. Regulation of beta 1- and beta 3-adrenergic agonist-stimulated lipolytic response in hyperthyroid and hypothyroid rat white adipocytes. Br J Pharmacol. 2000 Feb;129(3):448-56. doi: 10.1038/sj.bjp.0703008. PMID 10711342
- [Background] Mentuccia D, Proietti-Pannunzi L, Tanner K, Bacci V, Pollin TI, Poehlman ET, Shuldiner AR, Celi FS. Association between a novel variant of the human type 2 deiodinase gene Thr92Ala and insulin resistance: evidence of interaction with the Trp64Arg variant of the beta-3-adrenergic receptor. Diabetes. 2002 Mar;51(3):880-3. doi: 10.2337/diabetes.51.3.880. PMID 11872697